CLINICAL TRIAL: NCT01060969
Title: Tadalafil and Acetazolamide Versus Acetazolamide in Acute Mountain Sickness Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Head of the Center for Travel and Geographic Medicine, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-07-3977-ES-CTIL
Record Dates: First submitted 2008-11-03; First posted 2010-02-02 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Pulmonary Edema; Cerebral Edema
Keywords: Acute Mountain Sickness; travellers; Acetazolamide; Tadalafil; Acute Mountain Sickness assessed by Lake Louise score; High altitude pulmonary edema; High altitude cerebral edema
MeSH Terms: conditions — Pulmonary Edema; Brain Edema; Altitude Sickness | interventions — Tadalafil; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Active Comparator): acetazolamide 125 mg BID
  Interventions: Drug: Acetazolamide
- Acetazolamide and Tadalafil (Experimental): Intervention arm
  Interventions: Drug: Tadalafil and acetazolamide

INTERVENTIONS:
Drug: Tadalafil and acetazolamide — Experimental arm: Tadalafil 20 mg daily + acetazolamide 125 mg BID beginning above 3000 m altitude.
  Arms: Acetazolamide and Tadalafil
Drug: Acetazolamide — Active comparator arm (control): acetazolamide 125 mg BID beginning above 3000 m altitude
  Arms: Acetazolamide

SUMMARY:
To evaluate the additive value of tadalafil given together with Diamox (acetazolamide) in preventing acute mountain sickness in travelers to high altitude areas.

DETAILED DESCRIPTION:
A randomized controlled study comparing:

Tadalafil [20mg x1/day] and acetazolamide [125mg x2 day], versus Acetazolamide [125mg x2 day] alone, in trekkers to altitude > 3,000 m.

ELIGIBILITY:
Inclusion Criteria:

* Participant in trekking to high altitude
* Agreement to sign the informed consent.

Exclusion Criteria:

* No agreement to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Results will be evaluated by using the Lake Louise AMS scoring system | one month after travel

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Center of Geographic Medicine, Tel Litwinsky
  - Sheba Medical Ctr., Tel Litwinsky
  - Tel Litwinsky

REFERENCES:
- [Result] Leshem E, Caine Y, Rosenberg E, Maaravi Y, Hermesh H, Schwartz E. Tadalafil and acetazolamide versus acetazolamide for the prevention of severe high-altitude illness. J Travel Med. 2012 Sep-Oct;19(5):308-10. doi: 10.1111/j.1708-8305.2012.00636.x. Epub 2012 Jul 30. PMID 22943271